CLINICAL TRIAL: NCT05190783
Title: Partial Versus Complete Pulpotomy Using Three Different Materials in Primary Molars: a Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVCPUTDMIPMACS
Record Dates: First submitted 2021-12-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2019-02

CONDITIONS: Decayed Primary Molars
Keywords: Partial Pulpotomy; pulpotomy; MTA; Theracal; Formocresol
MeSH Terms: interventions — formocresol; Pemetrexed; mineral trioxide aggregate; TheraCal; Pulpotomy

STUDY DESIGN:
Who Masked: Participant
Masking Description: the children and their parents are blinded from the material that will be used and the technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- formocresol pulpotomy (Experimental): gold standard arm which pulpotomy will be done with formocresol
  Interventions: Drug: Formocresol; Procedure: pulpotomy
- formocresol partial pulpotomy (Active Comparator): partial pulpotomy will be done with formocresol
  Interventions: Drug: Formocresol; Procedure: partial pulpotomy
- MTA pulpotomy (Active Comparator): in this group complete pulpotomy will be done with MTA
  Interventions: Drug: MTA; Procedure: pulpotomy
- MTA partial pulpotomy (Active Comparator): in this study group partial pulpotomy will be done with MTA
  Interventions: Drug: MTA; Procedure: partial pulpotomy
- pulpotomy with Theracal LC (Active Comparator): in this study group complete pulpotomy will be done with Theracal LC
  Interventions: Drug: TheraCal; Procedure: pulpotomy
- partial pulpotomy with Theracal LC (Active Comparator): in this study group partial pulpotomy technique will be done with Theracal LC
  Interventions: Drug: TheraCal; Procedure: partial pulpotomy

INTERVENTIONS:
Drug: Formocresol — mixture of formalin, cresol and glycerine used for fixation of pulp tissues
  Arms: formocresol partial pulpotomy; formocresol pulpotomy
Drug: MTA — material used for pulp regeneration, direct and indirect pulp capping
  Other Names: Mineral trioxide aggregate
  Arms: MTA partial pulpotomy; MTA pulpotomy
Drug: TheraCal — light cured resin modified calcium silicate filled liner designed for use in direct and indirect pulp capping
  Arms: partial pulpotomy with Theracal LC; pulpotomy with Theracal LC
Procedure: pulpotomy — removal of the carious tooth structure and unroofing of the pulp chamber with a round carbide bur with high speed and water spray. The coronal pulp tissue will be then removed using a #4 carbide bur with slow speed and sharp spoon excavator.
  Arms: MTA pulpotomy; formocresol pulpotomy; pulpotomy with Theracal LC
Procedure: partial pulpotomy — complete removal of caries till exposure occurs. The exposed surface of the pulp will be gently removed using a sterile round diamond bur and a high-speed, water-cooled handpiece with light hand pressure. The removal of the pulp did not exceed approximately two mm.
  Arms: MTA partial pulpotomy; formocresol partial pulpotomy; partial pulpotomy with Theracal LC

SUMMARY:
The purposes of the study to compare partial pulpotomy versus complete pulpotomy in primary molars using three different materials (Formocresol, MTA, Theracal LC) . After 6, 9, 12 and 15 months follow up each case will be evaluated radiographically and clinically. the radiographic criteria to be evaluated are (radiolucency, resorption, widening in periodontal ligament space, Crypt involvement) and clinical criteria are ( pain, tenderness, fistula, abnormal mobility) upon these criteria some recommendations will be made on success and failure rate of each material and each technique.

DETAILED DESCRIPTION:
In children, deep carious lesions represent the most common disease of primary teeth; 42% of children aged 2 to 11 have dental carious lesions in their primary teeth, with an average of 1.6 decayed teeth per child. The most important objective of pediatric dentistry treatment is the preservation of functional primary teeth until natural exfoliation. In the era of conservative dentistry we are now focusing on repair rather than replacement.

Challenges regarding the best treatment modality in primary molars with deep carious lesions that are free of signs or symptoms have continued over the years. Based on a recent systematic review and a new American Academy of Pediatric Dentistry (AAPD) Guideline for vital pulp therapy in primary teeth, indirect pulp therapy (IPT), direct pulp cap (DPC), and pulpotomy are all viable options for treating the pulp in primary teeth with deep carious lesions.

Partial pulpotomy (PP) was originally a means of preserving the remaining coronal and radicular pulp tissues in permanent teeth after a traumatic pulp exposure. In 1982, Cvek introduced this technique for permanent traumatized teeth with complicated crown fracture, which involved removing two mm of pulp and then dressing the non-inflamed pulp with calcium hydroxide. However, according to the new AAPD best practices recommendation, PP is also indicated in young permanent teeth with a carious pulp exposure in which pulpal bleeding can be controlled within several minutes.

Calcium Hydroxide PP of primary molar teeth with deep carious lesions is used in studies conducted by Schroder and Trairatvorakul. Schroder. showed that the clinical-radiographic success rate of primary molar teeth one year after PP was 83 percent; they concluded that PP has the same favorable outcome as cervical formocresol pulpotomy (FP).

If the pulp is diagnosed as normal or as having reversible pulpitis, a new regenerative material is recommended as the dressing material. In comparison with complete pulpotomy (i.e., removal of the entire pulp chamber), PP has several advantages; it causes limited injury to the pulp and limited loss of tooth substances, and this is important for pulpal healing and easier restoration.

Pulpotomy is the pulp treatment most commonly used for primary teeth with a deep carious lesion approaching the pulp. With pulpotomy, a portion of the pulp is removed: the coronal pulp is removed and the radicular pulp is preserved. After treatment, the cavity is filled with a medicament followed by a final restoration.

Formocresol pulpotomy (FCP) was developed in 1932 by Charles A. Sweet.". The original FCP was a three-appointment procedure which has been reduced to a one-appointment procedure; it is still the most common treatment for primary teeth with caries approaching the pulp.

Studies have shown formocresol therapy to have a success rate between 70% and 90%.Histologic results have been variable in contrast to the high clinical success rate. Formocresol is still considered a gold standard by which all new modalities are compared.

MTA is used in pulp capping whether indirect or directly it has the advantage of biocompatibility to the pulp tissues and stimulates the odontoblast for thicker secondary dentine formation without tunnel defects and formation of hydroxyapatite like material to seal the pulp tissues. Although it has slow setting time, discolor the tooth, relatively high cost compared to the gold stander calcium hydroxide.

TheraCal light Cured (LC) is a single paste calcium silicate-based material promoted by the manufacturer for use as a pulp capping agent and as a protective liner for use with restorative materials, cement, or other base materials. The material might be very likable for clinicians because of its ease of handling. According to Alberto Danga in 2009 the cytotoxic effect of resin-based light-cured (Theracal) on human pulp tissue was least when compared to other materials.

There is a lack of evidence in partial pulpotomy treating primary teeth. In this study a Randomized control trial will be performed to have an evidence based answer for treating primary teeth with partial pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

* No history of spontaneous or nocturnal pain.
* History of transient pain of sensitivity resulting from various stimuli: hot, cold and sweets.
* Patient who had a bilateral deep carious lesion at second primary molars.
* absence of tenderness to percussion
* absence of physiologic or pathologic tooth mobility
* Radiographic evidence of no internal or external resorption.
* There is not an intraradicular or periapical bone loss or widening of the periodontal ligament space.

Exclusion Criteria:

* history of spontaneous or nocturnal pain.
* Patient who had a unilateral deep carious lesion.
* presence of tenderness to percussion
* presence of physiologic or pathologic tooth mobility
* Radiographic evidence of internal or external resorption.
* There is an intraradicular or periapical bone loss or widening of the periodontal ligament space.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
post operative pain | 15 months
  numerical/visual analogue scale 0 no pain 10 worst possible pain

SECONDARY OUTCOMES:
radiolucency | 15 months
  measuring tool is periapical xray
fistula | 15 months
  visual inspection
tooth mobility | 15 months
  clinical method of assessing tooth mobility 0 no mobility 3 mobility more than 2 mm bucco-lingualy
tenderness | 15 months
  percussion test with numerical/visual analogue scale 0 no pain 10 worst possible pain
root resorption | 15 months
  periapical xray
widening in periodontal ligament space | 15 months
  periapical xray
permanent tooth crypt involvement | 15 months
  periapical xray

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planning to publish my paper on pediatric dental journals
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Smail-Faugeron V, Porot A, Muller-Bolla M, Courson F. Indirect pulp capping versus pulpotomy for treating deep carious lesions approaching the pulp in primary teeth: a systematic review. Eur J Paediatr Dent. 2016 Jun;17(2):107-12. PMID 27377108
- [Result] Katz CR, de Andrade Mdo R, Lira SS, Ramos Vieira EL, Heimer MV. The concepts of minimally invasive dentistry and its impact on clinical practice: a survey with a group of Brazilian professionals. Int Dent J. 2013 Apr;63(2):85-90. doi: 10.1111/idj.12018. Epub 2013 Mar 12. PMID 23550521
- [Result] Dhar V, Marghalani AA, Crystal YO, Kumar A, Ritwik P, Tulunoglu O, Graham L. Use of Vital Pulp Therapies in Primary Teeth with Deep Caries Lesions. Pediatr Dent. 2017 Sep 15;39(5):146-159. PMID 29070150
- [Result] Cvek M, Cleaton-Jones PE, Austin JC, Andreasen JO. Pulp reactions to exposure after experimental crown fractures or grinding in adult monkeys. J Endod. 1982 Sep;8(9):391-7. doi: 10.1016/S0099-2399(82)80092-7. No abstract available. PMID 6957533
- [Result] Schroder U, Szpringer-Nodzak M, Janicha J, Wacinska M, Budny J, Mlosek K. A one-year follow-up of partial pulpotomy and calcium hydroxide capping in primary molars. Endod Dent Traumatol. 1987 Dec;3(6):304-6. doi: 10.1111/j.1600-9657.1987.tb00639.x. No abstract available. PMID 3481571
- [Result] Parirokh M, Torabinejad M, Dummer PMH. Mineral trioxide aggregate and other bioactive endodontic cements: an updated overview - part I: vital pulp therapy. Int Endod J. 2018 Feb;51(2):177-205. doi: 10.1111/iej.12841. Epub 2017 Sep 21. PMID 28836288
- [Result] Camp JH. Diagnosis dilemmas in vital pulp therapy: treatment for the toothache is changing, especially in young, immature teeth. J Endod. 2008 Jul;34(7 Suppl):S6-12. doi: 10.1016/j.joen.2008.03.020. PMID 18565375
- [Result] Wunsch PB, Kuhnen MM, Best AM, Brickhouse TH. Retrospective Study of the Survival Rates of Indirect Pulp Therapy Versus Different Pulpotomy Medicaments. Pediatr Dent. 2016 Oct 15;38(5):406-411. PMID 28206897
- [Result] George V, Janardhanan SK, Varma B, Kumaran P, Xavier AM. Clinical and radiographic evaluation of indirect pulp treatment with MTA and calcium hydroxide in primary teeth (in-vivo study). J Indian Soc Pedod Prev Dent. 2015 Apr-Jun;33(2):104-10. doi: 10.4103/0970-4388.155118. PMID 25872627
- [Result] El Meligy OA, Allazzam S, Alamoudi NM. Comparison between biodentine and formocresol for pulpotomy of primary teeth: A randomized clinical trial. Quintessence Int. 2016;47(7):571-80. doi: 10.3290/j.qi.a36095. PMID 27175451
- [Result] Poggio C, Arciola CR, Beltrami R, Monaco A, Dagna A, Lombardini M, Visai L. Cytocompatibility and antibacterial properties of capping materials. ScientificWorldJournal. 2014;2014:181945. doi: 10.1155/2014/181945. Epub 2014 May 18. PMID 24959601